CLINICAL TRIAL: NCT01428375
Title: Evaluation of Intravenous Infusion of Paracetamol as Intrapartum Analgesic in the First Stage of Labor: a Double-blind Randomized Trial
Brief Title: Intravenous Infusion of Paracetamol for Intrapartum Analgesia of Labor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Elbohoty, Lecturer in OB GYN, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PARACETAMOL-INTRAPARTUM; PARACETAMOL-INTRAPARTUM (Other: Pharma Tech company)
Record Dates: First submitted 2011-08-15; First posted 2011-09-05 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Labor Pain
Keywords: intravenous paracetamol; intrapartum analgesia; labor pain; intrapartum pains
MeSH Terms: conditions — Labor Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (1) Active (Paracetamol) arm: n=60 (Active Comparator): (Paracetamol)
  Interventions: Drug: (1) Paracetamol injection
- (2) Placbo (Sterile water) arm: n=60 (Placebo Comparator): Sterile water
  Interventions: Other: Sterile water

INTERVENTIONS:
Drug: (1) Paracetamol injection — Drugs: (1) Bottle containing 1000 mg Paracetamol in 100 ml solution for intravenous infusion
  Arms: (1) Active (Paracetamol) arm: n=60
Other: Sterile water — Drugs: (2) Bottle containing 100 ml sterile water for intravenous infusion
  Arms: (2) Placbo (Sterile water) arm: n=60

SUMMARY:
This is a double-blind randomized trial evaluates the efficacy of intravenous infusion of Paracetamol as intrapartum analgesic in the first stage of labour.

DETAILED DESCRIPTION:
Comparison of efficacy and safety of intravenous infusion of paracetamol versus placebo (intravenous sterile water infusion) in parturient women in active first phase of labour and requiring intrapartum analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-35 years.
2. Primigravida.
3. The gestational age between 37- 42 weeks.
4. Patient seeking analgesia.
5. Single viable fetus.
6. Vertex presentation.
7. Spontaneous onset of labor.
8. 1st stage of labor with cervical dilatation 3-4 cm ( in active phase).

Exclusion Criteria:

1. Extreme of age (below 18-above 35).
2. Multiparity.
3. Multiple gestation.
4. Malpresentation.
5. Major degree of cephalopelvic disproportion.
6. Any medical disorder with pregnancy e.g., Rheumatic heart disease, Diabetes mellitus, Hypertension, Anemia.
7. Induction of labor.
8. Cervical dilatation exceeds exceeding 4 cm.
9. Use of any other kind of analgesia before recruitment in the study.
10. Scared uterus.
11. Fetal distress.
12. Antepartum hemorrhage.
13. Intrapartum bleeding.
14. Polyhydramnios.
15. Pre-mature rupture of membranes.
16. Intra uterine infections.
17. Hypersensitivity to paracetamol.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of intravenous infusion of paracetamol in comparison with placebo (sterile water for injection) in labouring women | Start of medication till end of first stage of labour. Participants will be followed for the duration of labour, an expected average of 8 hours.
  By recoding the need for a rescue additional analgesia and measuring the degree of pain relief (Visual analogue score) during the labor process.

SECONDARY OUTCOMES:
To document safety | Start of medication till delivery and neonatal assesment. Participants will be followed during this duration of labour, an expected average of 10 hours.
  By assessing the adverse events recorded during the study either maternal or fetal/neonatal.
To correlate with the duration of labor | Start of medication till end of second stage of labour. Participants will be followed for the duration of labour, an expected average of 9 hours.
  The difference between both groups regarding labour duration

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed E Elbohoty, MD, Principal Investigator — OB GYN Department, faculty of Medicine, ASU
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Abd-El-Maeboud KH, Elbohoty AE, Mohammed WE, Elgamel HM, Ali WA. Intravenous infusion of paracetamol for intrapartum analgesia. J Obstet Gynaecol Res. 2014 Nov;40(11):2152-7. doi: 10.1111/jog.12465. Epub 2014 Aug 11. PMID 25132459